CLINICAL TRIAL: NCT01371396
Title: Effect of Dietary Macronutrient Composition on Liver Substrate Metabolism
Brief Title: Effect of Dietary Macronutrient Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Elizabeth Parks, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 5RL-1DK081187
Record Dates: First submitted 2011-06-07; First posted 2011-06-10 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Metabolic Syndrome; Non-alcoholic Fatty Liver Disease; Obesity
Keywords: Metabolic syndrome; Non-alcoholic fatty liver disease; Obesity Metabolism; Stable isotopes; Dietary weight loss
MeSH Terms: conditions — Metabolic Syndrome; Non-alcoholic Fatty Liver Disease; Obesity | interventions — Diet, Fat-Restricted; Diet, Carbohydrate-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hispanic subjects (Other): Subjects will identify as Hispanic ethnicity.
  Interventions: Other: Low-fat diet; Other: Low-carbohydrate diet
- African American subjects (Other): Subjects will self-identify as African American in origin.
  Interventions: Other: Low-fat diet; Other: Low-carbohydrate diet

INTERVENTIONS:
Other: Low-fat diet — The subject will consume a diet that is calorically restricted to cause at least a 6% body weight loss over 4 months. Fat will make up less than 30% of dietary energy.
Other: Low-carbohydrate diet — The diet will be restricted in energy to cause at least a 6% loss of body weight over a 4 month period. Carbohydrate will provide less than 40% of total dietary energy.

SUMMARY:
The purpose of this study is to understand why Hispanics who are overweight have a higher incidence of fatty liver disease.

DETAILED DESCRIPTION:
Obesity is a major factor driving the increased prevalence of hepatic steatosis in the US. However, little is known regarding the relationship between dietary intake and hepatic fat deposition or about the factors that promote loss of hepatic steatosis. Here, the investigators will determine how differences in dietary composition affect the development and regression of fatty liver. The investigators hypothesize that Hispanic subjects with metabolic syndrome will have higher liver fat synthesis rates compared to African American subjects.

Using detailed in vivo, serial measurements of fuel metabolism (GC/MS and NMR) fatty acid metabolism will be measured in the liver and periphery. This will be the first study in which these two methodologies are used together to assess both glucose and fatty acid metabolism in the same subjects. Subjects will be tested before and after a dietary weight-loss intervention producing 6% body weight loss over 5 months.

The specific aims are as follows:

AIM 1: Determine the contribution of peripheral and dietary fat to liver-TG in Hispanics and African Americans with metabolic syndrome.

Hypothesis: De novo lipogenesis will contribute to liver-TG in greater quantities compared to African Americans.

AIM 2: Determine the effects of low-CHO and low-fat diets on liver fat regression.

Hypothesis: Compared to a low-fat diet, a low-CHO diet will markedly decrease markers of inflammation coincident with greater improvements in insulin sensitivity as assessed by an intravenous glucose tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* Elevated serum ALT or metabolic syndrome
* African American or Hispanic
* Nondiabetic
* Men or women
* Smokers and nonsmokers
* Pre- and post-menopausal (+/- HRT)
* Stable body weight
* Age 20-65 years
* BMI between 25-45 kg/m2

Exclusion Criteria:

* Diabetes or Pregnancy
* Ethanol intake: males > 140 g/week, females > 70 g/week
* Chronic hepatitis B or chronic hepatitis C
* Hemochromatosis or Wilson's Disease
* Autoimmune hepatitis or primary biliary cirrhosis

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-09-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
de novo lipogenesis | Change from Baseline in fatty acid synthesis at 5 months
  In vivo measurement is made of liver fatty acid synthesis using stable isotope administration and analysis of plasma samples by GS/MS

SECONDARY OUTCOMES:
Dietary fatty acid clearance to liver | Change from Baseline in dietary fat clearance at 5 months
  Using a dietary stable isotope we will quantitate fat absorption and recycling of fat through the liver.
Adipose fatty acid flux | Change from Baseline in adipose fat flux at 5 months
  A stable isotope is infused and the rate of adipose fatty acid release is calculated after analyzing blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Parks, PhD, Principal Investigator — UTSW Medical Center
Locations (1):
- Center for Human Nutrition, Dallas, Texas, United States

REFERENCES:
- [Result] Shetty S, Ramos-Roman MA, Cho YR, Brown J, Plutzky J, Muise ES, Horton JD, Scherer PE, Parks EJ. Enhanced fatty acid flux triggered by adiponectin overexpression. Endocrinology. 2012 Jan;153(1):113-22. doi: 10.1210/en.2011-1339. Epub 2011 Nov 1. PMID 22045665
- [Result] Ramos-Roman MA, Sweetman L, Valdez MJ, Parks EJ. Postprandial changes in plasma acylcarnitine concentrations as markers of fatty acid flux in overweight and obesity. Metabolism. 2012 Feb;61(2):202-12. doi: 10.1016/j.metabol.2011.06.008. Epub 2011 Aug 5. PMID 21820684
- [Result] Sunny NE, Parks EJ, Browning JD, Burgess SC. Excessive hepatic mitochondrial TCA cycle and gluconeogenesis in humans with nonalcoholic fatty liver disease. Cell Metab. 2011 Dec 7;14(6):804-10. doi: 10.1016/j.cmet.2011.11.004. PMID 22152305
- [Result] Satapati S, Kucejova B, Duarte JA, Fletcher JA, Reynolds L, Sunny NE, He T, Nair LA, Livingston KA, Fu X, Merritt ME, Sherry AD, Malloy CR, Shelton JM, Lambert J, Parks EJ, Corbin I, Magnuson MA, Browning JD, Burgess SC. Mitochondrial metabolism mediates oxidative stress and inflammation in fatty liver. J Clin Invest. 2016 Apr 1;126(4):1605. doi: 10.1172/JCI86695. Epub 2016 Apr 1. No abstract available. PMID 27035816
- [Result] Lee JJ, Lambert JE, Hovhannisyan Y, Ramos-Roman MA, Trombold JR, Wagner DA, Parks EJ. Palmitoleic acid is elevated in fatty liver disease and reflects hepatic lipogenesis. Am J Clin Nutr. 2015 Jan;101(1):34-43. doi: 10.3945/ajcn.114.092262. Epub 2014 Nov 19. PMID 25527748
- [Result] Lambert JE, Parks EJ. Getting the label in: practical research strategies for tracing dietary fat. Int J Obes Suppl. 2012 Dec;2(Suppl 2):S43-50. doi: 10.1038/ijosup.2012.22. Epub 2012 Dec 11. PMID 27152153
- [Derived] Lambert JE, Ramos-Roman MA, Valdez MJ, Browning JD, Rogers T, Parks EJ. Weight loss in MASLD restores the balance of liver fatty acid sources. J Clin Invest. 2025 May 1;135(9):e174233. doi: 10.1172/JCI174233. eCollection 2025 May 1. PMID 40309768
- [Derived] Ramos-Roman MA, Lapidot SA, Phair RD, Parks EJ. Insulin activation of plasma nonesterified fatty acid uptake in metabolic syndrome. Arterioscler Thromb Vasc Biol. 2012 Aug;32(8):1799-808. doi: 10.1161/ATVBAHA.112.250019. Epub 2012 Jun 21. PMID 22723441